CLINICAL TRIAL: NCT04499521
Title: A Randomized, Non-Inferiority Study of a Hydrogel Packing System Compared to Standard of Care Packing During Image-Guided High-Dose Rate Brachytherapy Boost for Cervical Cancer
Brief Title: A Randomized Study to Compare a Hydrogel Packing System to Standard Packing During HDR Brachytherapy for Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: BrachyFoam, LLC (Unknown)
Responsible Party: Principal Investigator, Kara Romano, MD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR 200128
Record Dates: First submitted 2020-07-22; First posted 2020-08-05 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer
Keywords: Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Both groups will have two fractions of brachytherapy with a standard packing system and two fractions of brachytherapy with BrachyGel VHPS - only the timing will be different between the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm A: BrachyGel in fractions 3 and 5 (Experimental): BrachyGel VHPS in fractions 3 and 5 and standard packing in fractions 2 and 4
  Interventions: Device: BrachyGel VHPS
- Arm B: BrachyGel in fractions 2 and 4 (Experimental): BrachyGel VHPS in fractions 2 and 4 and standard packing in fractions 3 and 5
  Interventions: Device: BrachyGel VHPS

INTERVENTIONS:
Device: BrachyGel VHPS — Packing system for administering brachytherapy in cervical cancer patients

SUMMARY:
In this study, a new, low cost packing system ("BrachyGel VHPS") is being tested as a packing option during brachytherapy along with standard options to make sure that it keeps the unrelated organs away from radiation at least as well as the standard options, and to better understand the safety and patient discomfort associated with BrachyGel VHPS and the standard packing options.

DETAILED DESCRIPTION:
As part of vaginal brachytherapy, the organs that do not need to receive radiation (unrelated organs) are moved out of the way of the radiation with a "packing system". The usual low cost and available standard of care packing systems to move these unrelated organs out of the way can sometimes be uncomfortable for the patient, may not move all of the unrelated organs all the way out of the radiation's path, and rely on the doctor to place them correctly.

If you participate, you will receive 5 fractions of brachytherapy according to standard clinical care. For three of the fractions, a standard packing option will be used and for two of them BrachyGel VHPS will be used. For the first fraction both groups will have the same packing option but participants will be randomized to either have BrachyGel during fractions 2 and 4 or during fractions 3 and 5. You'll be asked to complete a questionnaire after fractions 2-5 to get your feedback on any discomfort you have during or after brachytherapy from the packing system.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy showing cancer of the cervix (squamous cell carcinoma, adenocarcinoma, adenosquamous, neuroendocrine, etc)
2. FIGO IB1 - IVB Staging according to FIGO and TNM guidelines
3. Planning to receive brachytherapy as a part of the definitive treatment for cervical cancer
4. Karnofsky performance status (KPS) ≥ 70 or ECOG status ≤1
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Age ≥ 18 years
7. Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

1. History of pelvis or abdominal radiation therapy (RT) that is not a part of the definitive treatment plan for the cancer of interest"
2. History of total or partial hysterectomy
3. Plan to receive external beam RT (EBRT) alone as the definitive treatment plan for the cancer of interest
4. Known pregnancy or lactation (no pregnancy test required prior to participation)
5. Known contraindications to brachytherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Romano, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at one academic medical center between March 2021 and September 2022. Participants were randomized with equal allocation to each ordering (Arm A or Arm B) using a stratified block randomization scheme with varying block sizes (of 2-4). Randomization occurred prior to the 2nd fraction of brachytherapy.
Pre-assignment Details: Fraction 1 for all participants (both Arms) was performed with standard of care packing. One patient of the 21 patients enrolled and randomized did not receive brachytherapy due to disease progression.
Period: Overall Study
Arm/Group | Arm A: BrachyGel in Fractions 3 and 5 | Arm B: BrachyGel in Fractions 2 and 4
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: BrachyGel in Fractions 3 and 5 | Arm B: BrachyGel in Fractions 2 and 4 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 52.9 [34 to 71] | 51 [38 to 70] | 51.95 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Dosimetry Comparison of Packing System in OARs
Description: The mean difference in bladder and rectum doses between Gauze and BrachyGel for fractions 2 and 3
Time Frame: Fractions 2 and 3 about 1 - 2 weeks after starting brachytherapy
Population: 19 participants were evaluated. A major protocol deviation that occurred for one ARM B subject during fraction (Fx) 2 of brachytherapy (use of an incorrect packing method). This subject is not included in the analysis of this endpoint.
Measure: Mean (Standard Deviation); unit: Mean in Dose (Gray)
Groups:
- ARM A Fraction 2: Gauze
  ARM A: BrachyGel VHPS in fractions 3 and 5 and standard packing in fractions 2 and 4
- ARM A Fraction 3: BrachyGel
  ARM A: BrachyGel VHPS in fractions 3 and 5 and standard packing in fractions 2 and 4
- ARM B Fraction 2: BrachyGel
  ARM B: BrachyGel VHPS in fractions 2 and 4 and standard packing in fractions 3 and 5
- ARM B Fraction 3: Gauze
  ARM B: BrachyGel VHPS in fractions 2 and 4 and standard packing in fractions 3 and 5
Arm/Group | ARM A Fraction 2 | ARM A Fraction 3 | ARM B Fraction 2 | ARM B Fraction 3
Number analyzed (Participants) | 10 | 10 | 9 | 10
Mean in Dose (Gray)
  Bladder D2cc | 3.436 (0.684) | 3.319 (0.586) | 3.636 (0.772) | 3.573 (0.791)
  Rectum D2cc | 3.071 (0.386) | 3.26 (0.357) | 3.211 (0.693) | 3.03 (0.722)
  Bladder D1cc | 3.745 (0.774) | 3.601 (0.586) | 4.026 (0.845) | 3.908 (0.828)
  Rectum D1cc | 3.417 (0.492) | 3.591 (0.405) | 3.51 (0.789) | 3.316 (0.812)
  Bladder D0.1cc | 4.457 (1.035) | 4.311 (0.78) | 4.911 (1.018) | 4.705 (0.916)
  Rectum D0.1cc | 4.117 (0.713) | 4.34 (0.681) | 4.381 (1.06) | 4.028 (1.134)
  HR-CTVD90 | 6.518 (1.313) | 6.638 (0.901) | 5.917 (0.893) | 6.575 (0.869)
Statistical Analysis 1: Comparison: ARM A Fraction 2 vs ARM A Fraction 3; Mean difference between Gauze and Gel ARM A Bladder D2cc; Test type: Other; Median Difference (Final Values) = 0.12, 95% CI 2-sided [-0.27 to 0.50]
Statistical Analysis 2: Comparison: ARM B Fraction 2 vs ARM B Fraction 3; Mean difference between Gauze and Gel ARM B Bladder D2cc; Test type: Other; Median Difference (Final Values) = 0.01, 95% CI 2-sided [-0.94 to 0.96]
Statistical Analysis 3: Comparison: ARM A Fraction 2 vs ARM A Fraction 3; Mean difference between Gauze and Gel ARM A Rectum D2cc; Test type: Other; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.54 to 0.16]
Statistical Analysis 4: Comparison: ARM B Fraction 2 vs ARM B Fraction 3; Mean difference between Gauze and Gel ARM B Rectum D2cc; Test type: Other; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.67 to 0.29]

2. Secondary Outcome: Adverse Events
Description: Frequency and intensity (CTCAE v5 grade) of AEs
Time Frame: From the completion of the 2nd brachytherapy treatment to 1 month after the last brachytherapy treatment (up to 70 days)
Population: All participants who received at least Brachytherapy Fraction 2
Measure: Number; unit: Occurences
Groups:
- BrachyGel: A Research Packing system for administering brachytherapy in cervical cancer patients.
  AEs related to Brachygel
- Gauze: A Standard of care packing method for administering brachytherapy in cervical cancer patients.
  AEs related to Gauze
- Other: Not Related to either packing system
Arm/Group | BrachyGel | Gauze | Other
Number analyzed (Participants) | 20 | 20 | 20
Occurences
  Vaginal pain Grade 2 | 2 | 0 | 2
  Vaginal pain Grade 1 | 0 | 0 | 3
  Vaginal hemorrhage (Spotting) Grade 1 | 1 | 1 | 2
  Vaginal dryness (itching) Grade 1 | 0 | 0 | 1
  Vaginal inflammation Grade 1 | 0 | 1 | 1
  Vaginal inflammation Grade 2 | 0 | 0 | 1
  Dysuria Grade 1 | 0 | 0 | 1
  Dysuria Grade 2 | 0 | 0 | 1
  Urinary urgency Grade 1 | 0 | 0 | 1
  Pelvic Pain Grade 3 | 0 | 0 | 1
  Pelvic pain (abdominal cramping) Grade 2 | 0 | 0 | 2
  Pelvic pain (abdominal cramping) Grade 1 | 0 | 0 | 3
  Fatigue Grade 2 | 0 | 0 | 1
  Fatigue Grade 1 | 0 | 0 | 1
  Diarrhea Grade 1 | 0 | 0 | 1
  Constipation Grade 1 | 0 | 0 | 2
  Dyspareunia Grade 1 | 0 | 0 | 1
  Dermatitis Radiation Grade 2 | 0 | 0 | 2
  Dizziness Grade 2 | 0 | 0 | 1
  Nausea Grade 2 | 0 | 0 | 1
  Vomiting Grade 2 | 0 | 0 | 1
  Cough Grade 1 | 0 | 0 | 1
  Bloating Grade 1 | 0 | 0 | 1
  Bone Pain Grade 1 | 0 | 0 | 1
  Facial Pain Grade 1 | 0 | 0 | 1
  UTI Grade 2 | 0 | 0 | 1
  Infection (Scabies)* Grade 3 | 0 | 0 | 1
  Vaginal Infection Grade 1 | 0 | 0 | 1

3. Secondary Outcome: Dosimetry Comparison of Packing System in OARs
Description: The mean difference in bladder and rectum doses between Gauze and BrachyGel for fractions 2 through 5.
Time Frame: Fractions 2 and 5 about 1 - 4 weeks after starting brachytherapy
Population: A major protocol deviation that occurred for one ARM B subject during fraction (Fx) 2 of brachytherapy (use of an incorrect packing method). Two subjects one from ARM A and one from ARM B only received 4 fractions of treatment. These subjects are not included in the analysis of this endpoint.
Measure: Mean (Standard Deviation); unit: Mean in dose (Gray)
Groups:
- ARM A Fraction 4: Gauze
  ARM A: BrachyGel VHPS in fractions 3 and 5 and standard packing in fractions 2 and 4
- ARM A Fraction 5: BrachyGel
  ARM A: BrachyGel VHPS in fractions 3 and 5 and standard packing in fractions 2 and 4
- ARM B Fraction 4: BrachyGel
  ARM B: BrachyGel VHPS in fractions 2 and 4 and standard packing in fractions 3 and 5
- ARM B Fraction 5: Gauze
  ARM B: BrachyGel VHPS in fractions 2 and 4 and standard packing in fractions 3 and 5
Arm/Group | ARM A Fraction 2 | ARM A Fraction 3 | ARM A Fraction 4 | ARM A Fraction 5 | ARM B Fraction 2 | ARM B Fraction 3 | ARM B Fraction 4 | ARM B Fraction 5
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 10 | 10 | 9
Mean in dose (Gray)
  Bladder D2cc | 3.436 (0.684) | 3.319 (0.586) | 3.287 (1.058) | 3.798 (0.771) | 3.636 (0.772) | 3.573 (0.791) | 3.157 (1.174) | 3.649 (0.916)
  Rectum D2cc | 3.071 (0.386) | 3.26 (0.357) | 3.035 (0.627) | 2.936 (0.847) | 3.211 (0.693) | 3.03 (0.722) | 2.761 (0.664) | 2.993 (0.67)
  Bladder D1cc | 3.745 (0.774) | 3.601 (0.586) | 3.611 (1.142) | 4.166 (0.873) | 4.026 (0.845) | 3.908 (0.828) | 3.453 (1.234) | 4.072 (0.977)
  Rectum D1cc | 3.417 (0.492) | 3.591 (0.405) | 3.378 (0.664) | 3.201 (0.919) | 3.51 (0.789) | 3.316 (0.812) | 3.015 (0.725) | 3.236 (0.73)
  Bladder D0.1cc | 4.457 (1.035) | 4.311 (0.78) | 4.322 (1.352) | 4.974 (1.144) | 4.911 (1.018) | 4.705 (0.916) | 4.287 (1.518) | 5.031 (1.186)
  Rectum D0.1cc | 4.117 (0.713) | 4.34 (0.681) | 4.2 (0.795) | 3.846 (1.054) | 4.381 (1.06) | 4.028 (1.134) | 3.817 (1.068) | 3.823 (0.835)
  HR-CTVD90 | 6.518 (1.313) | 6.638 (0.901) | 6.749 (1.501) | 6.692 (0.522) | 5.917 (0.893) | 6.575 (0.869) | 6.807 (1.262) | 6.284 (0.543)

ADVERSE EVENTS:
Time Frame: From completion of the 2nd brachytherapy treatment to 1 month after the last brachytherapy treatment (up to 70 days)
Description: Adverse events were not collected before the 2nd brachytherapy treatment. The 1st brachytherapy treatment is considered a part of baseline and was performed using gauze per standard of care for all subjects. The time from informed consent to 2nd brachytherapy was up to 14 days and the time from 1st brachytherapy to 2nd brachytherapy was up to 12 days.
Groups:
- BrachyGel for Arm A: Event occurred on or after the day BrachyGel VHPS was used on participants assigned to ARM A
  ARM A: Brachygel used during fractions 3 and 5 and standard packing in fractions 2 and 4
- Gauze for Arm A: Event occurred on or after the day Gauze was used on participants assigned to ARM A
  ARM A: Brachygel used during fractions 3 and 5 and standard packing in fractions 2 and 4
- Other for Arm A: Not associated with either packing system due the start date of the event (i.e. started during follow up).
  ARM A: Brachygel used during fractions 3 and 5 and standard packing in fractions 2 and 4
- BrachyGel for Arm B: Associated with BrachyGel VHPS for participants assigned to ARM B
  ARM B: Brachygel used during fractions 2 and 4 and standard packing in fractions 3 and 5
- Gauze for Arm B: Event occurred on or after the day Gauze was used on participants assigned to ARM B
  ARM B: Brachygel used during fractions 2 and 4 and standard packing in fractions 3 and 5
- Other for Arm B: Not associated with either packing system due the start date of the event (i.e. started during follow up).
  ARM B: Brachygel used during fractions 2 and 4 and standard packing in fractions 3 and 5
Arm/Group | BrachyGel for Arm A | Gauze for Arm A | Other for Arm A | BrachyGel for Arm B | Gauze for Arm B | Other for Arm B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10 | 5/10 | 5/10 | 3/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BrachyGel for Arm A (N=10) | Gauze for Arm A (N=10) | Other for Arm A (N=10) | BrachyGel for Arm B (N=10) | Gauze for Arm B (N=10) | Other for Arm B (N=10)
Vaginal Pain (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Vaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal Inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UTI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Scabies) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations of this study include unblinded participants, lack of MRI for treatment planning, and a smaller than planned sample size. The study was designed as a non-inferiority trial with a planned accrual of 40 participants (20 per arm); however, the trial accrued 20 participants. No formal statistical significance calculations were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT04499521/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT04499521/ICF_001.pdf